CLINICAL TRIAL: NCT02762123
Title: Effects of Concomitant Administration of BMS-986142 on the Single-dose Pharmacokinetics of Probe Substrates for CYP2C8, CYP2C9, CYP2C19, CYP3A4, and P-gp in Healthy Subjects
Brief Title: A Study to Assess the Effect of BMS-986142 on Pharmacokinetics (PK) of Probe Substrates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IM006-031
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — montelukast; Flurbiprofen; Omeprazole; Midazolam; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (BMS-986142: 200 mg) (Experimental): 200mg BMS-986142 administered orally once daily on specified days.
  Interventions: Drug: BMS-986142 200mg; Drug: BMS Drug-drug interaction cocktail (montelukast, flurbiprofen, omeprazole, midazolam, and digoxin)
- Cohort 2 (BMS-986142: 350 mg) (Experimental): 350mg BMS-986142 administered orally once daily on specified days.
  Interventions: Drug: BMS Drug-drug interaction cocktail (montelukast, flurbiprofen, omeprazole, midazolam, and digoxin); Drug: BMS-986142 350mg

INTERVENTIONS:
Drug: BMS-986142 200mg
  Arms: Cohort 1 (BMS-986142: 200 mg)
Drug: BMS Drug-drug interaction cocktail (montelukast, flurbiprofen, omeprazole, midazolam, and digoxin)
Drug: BMS-986142 350mg
  Arms: Cohort 2 (BMS-986142: 350 mg)

SUMMARY:
The study is being conducted to assess the effect of BMS-986142 on the single-dose PK parameters of montelukast, flurbiprofen, omeprazole, midazolam, and digoxin, probe drugs for (cytochome P450) CYP2C8, CYP2C9, CYP2C19, CYP3A4, and P-glycoprotein (P-gp), respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Target population: Healthy (current non-smokers) subjects as determined by medical history, surgical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory determinations.
3. Subjects with body mass index of 18 to 32 kg/m2, inclusive
4. Men, and women of nonchildbearing potential. Women must have documented proof that they are not of childbearing potential and must not be breastfeeding.
5. Males who are sexually active with women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of the study drug (3 days) plus 90 days (duration of sperm turnover) for a total of 93 days (approximately 14 weeks) after treatment completion. Female partners of male subjects are expected to use one of the highly effective methods of contraception listed in the protocol.

Exclusion Criteria:

1. History of any chronic or acute illness, recent infection, gastrointestinal disease, smoking and alcohol abuse, any significant drug allergy or allergy to digoxin, flurbiprofen, midazolam, omeprazole, or montelukast, Bruton's tyrosine kinase (BTK) inhibitors, immunologic or related compounds.
2. History of billiary disorder, asthma, bleeding disorder, cancer
3. Received live vaccine during last 12 weeks, active tuberculosis (TB) in last 3 years
4. Medical history indicative of an increased risk of arrhythmia.
5. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of montelukast, flurbiprofen, omeprazole, midazolam, and digoxin. | 57 samples up to day 26
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T))of montelukast, flurbiprofen, omeprazole, midazolam, and digoxin | 57 samples up to day 26
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of montelukast, flurbiprofen, omeprazole, midazolam, and digoxin | 57 samples up to day 26

SECONDARY OUTCOMES:
Safety endpoints include the incidence of adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation, and death | Days 1-26; for SAEs up to 30 days post discontinuation of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States

REFERENCES:
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx